CLINICAL TRIAL: NCT04244617
Title: Peer-supported Internet Mediated Psychological Treatment for Adults With Anxiety Disorders in Primary Care
Brief Title: Peer-supported Internet Mediated Psychological Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Drn EPN: 845-18
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Psychological Phenomena and Processes; Behavior and Behavior Mechanisms; Mental Disorder; Behavioral Disciplines and Activities
Keywords: iCBT; Primary Care; Anxiety; Drop-out; Peer-support; Mixed method design
MeSH Terms: conditions — Behavior; Mental Disorders; Motor Activity; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study is a mixed methods design consisting of an un-controlled pragmatic effectiveness study combined with semi-structured interviews
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iCBT with addition of peer-support (iCBT-PS) (Experimental): Participants in the iCBT-PS, are guided by both a psychologist and a peer-support in the iCBT-program used in the study.
  Interventions: Behavioral: iCBT with addition of peer-support

INTERVENTIONS:
Behavioral: iCBT with addition of peer-support — Peer-supporters and participants, as well as psychologists and participants, interact in the treatment program via asynchronous secure messages. Peer-supporters are able to give support and feedback on exercises. A reconciliation call via telephone is entered into the middle of the treatment and a follow-up call after completion of treatment conducted by the peer-support. The interaction between peer-supporters and participants is tracked by the psychologist.

SUMMARY:
This study evaluates the effect and experience of peer-support in internet mediated ACT (Acceptance and Commitment therapy) in an explorative pilot study with mixed method design conducted in primary care. Peer-supporters are certified support persons with personal experience of mental health problems and the process of rehabilitation, which becomes professionally active in care and support to patients in their recovery

DETAILED DESCRIPTION:
The study is a mixed methods design consisting of an un-controlled pragmatic effectiveness study combined with semi-structured interviews in order to investigate the participant´s experience of treatment. Participants were recruited from patients who were referred to a central unit for internet- CBT (Cognitive Behavioral therapy) in primary care in Västra Götaland region, Sweden. Peer-supporters were recruited through a swedish patient organization. Participants were adults 18 years of age or older with an anxiety disorder.

All participants were interviewed by a psychologist with a diagnostic instrument, a structured interview called PRIME-MD, before starting treatment. After the interview, all patients who were offered iCBT and met the inclusion criteria were requested to participate in the study.

Patients who accepted inclusion were guided by both a psychologist and a peer-support in the iCBT treatment used in the study. The iCBT treatment program used is a transdiagnostic program aimed at treating people with mild to moderate anxiety problems.

Quantitative data about psychosocial symptoms were collected, and qualitative data about the participants experience of treatment were collected through semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* participants must have reached the age of 18
* have access to a computer with internet Connection
* speak and understand Swedish
* meet the diagnostic criteria for an anxiety disorder (social anxiety, GAD, panic disorder, obsessive-compulsive disorder, or unspecified anxiety disorder).

Exclusion Criteria:

* have started medication or have made major changes regarding their medication in the past few months
* have serious suicidal ideation or suicide plans
* are expected to have complex problems or be in need of other care
* are under any other psychological treatment during the time of the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety symptoms | Baseline (Pre-treatment), post treatment (after 8 weeks) and by 3 month follow up
  Anxiety is measured with the GAD-7 instrument (Generalized Anxiety Disorder 7 item scale). The scale consists of 7 items. The score ranges from 0 to 21, with higher scores indicating more anxiety symptoms. There are thresholds for mild, medium and severe anxiety (Spitzer, Kroenke, Williams & Löwe 2006).
Change in Depressive symptoms | Baseline (Pre-treatment), post treatment (after 8 weeks) and by 3 month follow up
  Symptoms of depression is measured with Madrs-s (Montgomery Åsberg Depression Rating Scale; Montgomery & Åsberg, 1979). The instrument consists of 9 items. Scores ranges from 0 to 60, with higher scores indicating more depressive symptoms. There are cut-off points for symptom severity.
Change in symptoms of psychological distress | Baseline (Pre-treatment) and post treatment (after 8 weeks) (Since this instrument is provided in connection with the modules in the treatment program
  Symptoms of psychological distress is measured with the CORE-10 (Barkham et al., 2012). Score ranges from 0 to 40, with higher scores indicating more psychological distress. The instrument consists of 10 items and has clinical cut-off scores for general psychological distress.
Changes in feelings of empowerment | Baseline (Pre-treatment), post treatment (after 8 weeks) and by 3 month follow up
  Empowerment is measured with the Empowerment Scale (Rogers, Chamberlin, Ellison & Crean, 1997). The scale consists of 28 items which are answered on a four-point likert scale. Score ranges between 28 and 112. Higher scores indicates that the person feels more empowered.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Weineland, PhD, Study Chair — Department of psychology, University of Gothenburg, Sweden
Locations (1):
- Närhälsan, Primary care, Borås, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We will share the data if a corresponding author or otherwise authorized person asks for it
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code